CLINICAL TRIAL: NCT07376499
Title: Prospective, Single-arm, Phase II Clinical Study of Irinotecan Hydrochloride Liposome Injection Combined With Platinum and Immune Checkpoint Inhibitors Combined With Anlotinib for the Maintenance of Extensive Small Cell Lung Cancer After First-line Induction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Xiujuan Qu, professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-SCLC-LN01
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-04

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; liposome irinotecan; platinum; immune checkpoint inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Platinum; anlotinib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Irinotecan hydrochloride liposome injection combined with platinum and tislelizumab therapy in a 3-week treatment cycle , 4 cycles
  Interventions: Drug: Liposome Irinotecan; Drug: Platinum; Drug: Anlotinib; Drug: Toripalimab

INTERVENTIONS:
Drug: Liposome Irinotecan — Liposome irinotecan(50mg/m^2) will be administered by intravenous infusion on day 1 in a 3-week treatment cycle
Drug: Platinum — Carboplatin (AUC 4-5) or Cisplatin (60mg/m^2) will be administered by intravenous infusion on day 1 in a 3 week treatment cycle
Drug: Anlotinib — Anlotinib (8mg) will be administered orally in a 3-week treatment cycle, once a day from day 1 to day 14 of each cycle
Drug: Toripalimab — Toripalimab (240mg) will be administered by intravenous infusion on day 1 in a 3-week treatment cycle

SUMMARY:
To evaluate the efficacy and safety of liposome irinotecan combined with platinum and immune checkpoint inhibitor combined with antirotinib maintenance therapy after first-line induction

DETAILED DESCRIPTION:
1. Irinotecan hydrochloride liposome injection combined with platinum and tislelizumab therapy in a 3-week treatment cycle , 4 cycles Drug: Liposome irinotecan(50mg/m^2) will be administered by intravenous infusion on day 1 in a 3-week treatment cycle Drug: Carboplatin (AUC 4-5) or Cisplatin (60mg/m^2) will be administered by intravenous infusion on day 1 in a 3-week treatment cycle Drug: Toripalimab (240mg) will be administered by intravenous infusion on day 1 in a 3 week treatment cycle
2. Maintenance treatment, to disease progression or AE Drug: Toripalimab (240mg) will be administered by intravenous infusion on day 1 in a 3 week treatment cycle Drug: Anlotinib (8mg) will be administered orally in a 3-week treatment cycle, once a day from day 1 to day 14 of each cycle

ELIGIBILITY:
Inclusion Criteria:

* 1. Volunteer to join the study, sign the informed consent and sign the date, have good compliance, and cooperate with follow-up 2. Age≥18 years 3. Diagnosis of extensive stage small cell lung cancer (ES-SCLC) confirmed histologically or pathologically (according to American Veterans Lung Cancer Association, VALG staging) 4. ECOG 0-2 5. Subjects had not received any systemic treatment for ES-SCLC in the past (including chemotherapy, use of similar VEGFR inhibitors and immune checkpoint inhibitors, etc.) 6. Subjects with limited-stage small cell lung cancer (LS-SCLC) have received radiotherapy, chemotherapy, or chemoradiotherapy for more than 6 months 7. Expected survival ≥ 3 months 8. Must have measurable target lesions that meet RECIST1.1 criteria (CT scan length of tumor lesion >10mm); In patients with initial asymptomatic brain metastases, craniocerebral radiotherapy may be performed during induction chemotherapy 9. If the major organs are functioning normally, the following criteria are met:

  1. Blood routine examination must meet (no blood transfusion within 14 days, no hematopoietic factor and no drug correction) : ANC ≥ 1.5×10^9/L; HB ≥ 90 g/L; PLT ≥ 100×10^9/L
  2. Biochemical examination must meet the following criteria: TBIL ≤ 1.5ULN; ALT and AST≤ 2.5ULN;
  3. Renal function must meet the following criteria: serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥40 mL/min (using the standard Cockcroft-Gault formula)
  4. Coagulation function must meet: INR≤1.5 and APTT≤1.5ULN 10. Female who are fertile must have a serum or urine pregnancy test within 72 hours before the first medication and the result is negative. Fertile female and male subjects whose partners are fertile female must agree to a highly effective method of avoiding and breastfeeding during the study period until 90 days after the last dose of the study drug. The investigator or designee, in consultation with the subject, shall confirm that the subject understands the proper and consistent use of contraceptive methods 11. For males, they should be surgically sterilized or consent to a highly effective method of avoidance during the trial and for 90 days after the last administration of the experimental drug 12. Female participants had to agree not to breastfeed during the study period or for 180 days after the last dose of study treatment

Exclusion Criteria:

* 1. Patients with meningeal metastases or symptomatic brain metastases 2. Previous T cell co-stimulation or immune checkpoint therapy, including but not limited to cytotoxic T lymphocyte-associated antigen-4 (CTLA-4)inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, CD137 agonists, or other targeting T cell drugs; 3. Past treatment with anlotinib 4. Factors affecting oral medication, such as inability to swallow, post-GI resection, chronic diarrhea, intestinal obstruction, etc 5. Uncontrollable pleural effusion or ascites 6. Have any active autoimmune disease or history of autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (may be included after hormone replacement therapy), tuberculosis); Patients with skin conditions (such as vitiligo, psoriasis, or alopecia) that have been in complete remission from childhood asthma and do not require any intervention in adulthood and do not require systemic treatment may be included. Patients who require medical intervention with bronchodilators may not be included 7. Patients with congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500IU/ml), hepatitis C (HCV antibody positive and HCV-RNA above the lower detection limit of analytical methods), or co-infection with hepatitis B and hepatitis C 8. Urine routine suggests urinary protein ≥(++), or 24h urinary protein ≥2g or severe hepatic and renal insufficiency 9. Patients requiring systemic therapy with corticosteroids (>10mg/ day of prednisone or equivalent) or other immunosuppressants within 14 days prior to initial medication. In the absence of active autoimmune disease, inhaled or topical corticosteroids are permitted, as well as adrenal hormone replacement therapy at doses >10 mg/ day of prednisone efficacy 10. Patients who have been treated with anti-tumor vaccine or other immunostimulating anti-tumor agents (interferon, interleukin, thymosin, immunocell therapy, etc.) within 1 month prior to initial medication 11. Other malignant neoplasms were present within 5 years prior to admission, except for adequately treatable carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery 12. There is evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia, radiologically proven active pneumonia, and severe impairment of lung function 13. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90mmHg, despite optimal medical treatment 14. Patients with grade II or higher myocardial ischemia or myocardial infarction and poorly controlled arrhythmias (including QTc interval

  * 450ms in men and ≥470ms in women). According to the NYHA criteria, patients with grade III to # cardiac insufficiency, or those with left ventricular ejection fraction (LVEF) < 50% indicated by color Doppler ultrasound had myocardial infarction in the 6 months prior to enrollment, heart failure of New York Heart Society grade II or above, uncontrolled angina, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, and myocardial infarction. Or electrocardiogram suggests acute ischemia or abnormal active conduction system 15. Concurrent severe infection within 4 weeks prior to first dosing, or unexplained fever >38.5°C during screening/prior to first dosing 16. Major surgery, open biopsy, or significant trauma were performed within 28 days prior to enrollment 17. Aortic/venous thrombosis occurred within 6 months 18. The researchers assessed possible risk of severe hemoptysis, bleeding events, or wearing 19.Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation 20.Pregnant or lactating women; Fertile patients who are unwilling or unable to use effective contraception 21.Allergic reaction to any investigational drug or its ingredients 22.Any condition that the investigator believes is likely to harm the subject or cause the subject to be unable to meet or perform the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) To evaluate the efficacy of anti-tumor | baseline up to approximately 6 months

SECONDARY OUTCOMES:
Objective response rate (ORR) To evaluate the efficacy of anti-tumor | baseline up to approximately 6 months
Disease Control Rate (DCR) To evaluate the efficacy of anti-tumor | baseline up to approximately 6 months
overall survival (OS) To evaluate the efficacy of anti-tumor | baseline up to approximately 12 months
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] To identify the incidence of AE and SAE in clinical trial | From the initiation of the first dose to 14 days after the last dose